CLINICAL TRIAL: NCT05047900
Title: The Impact of SARS-CoV-2 Rapid Antigen Testing Kit Screening in Bangkok Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Yuvabadhana foundation (Unknown); Zero COVID Thailand (Unknown); Chulalongkorn University (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, Gasit Saksirisampant, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: COA. MURA2021/711
Record Dates: First submitted 2021-09-06; First posted 2021-09-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Covid19; SARS-CoV-2; Community Transmissions; Coronavirus Infections
Keywords: ATK; Covid19; Rapid antigen testing kit; Screening; Community transmissions; SARS-CoV-2; Coronavirus; Infectious diseases
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Communicable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rapid antigen testing kit use once weekly (Experimental): Community will use rapid antigen testing kit once weekly every Monday and will be asked to conduct a weekly self-test for 3 weeks.
  This research use COVID-19 Saliva Antigen Rapid Test from Tigsun COVID-19 Speichel Antigen-Schnelltest from Beijing Tigsun Diagnostics
  Interventions: Diagnostic Test: Rapid antigen testing kit
- Rapid antigen testing kit use twice weekly (Experimental): Community will use rapid antigen testing kit twice weekly every Monday and Thursday and will be asked to conduct a twice-weekly self-test for 3 weeks This research use COVID-19 Saliva Antigen Rapid Test from Tigsun COVID-19 Speichel Antigen-Schnelltest from Beijing Tigsun Diagnostics
  Interventions: Diagnostic Test: Rapid antigen testing kit
- Control (No Intervention): Did not routinely use Rapid antigen testing kit

INTERVENTIONS:
Diagnostic Test: Rapid antigen testing kit — COVID-19 Saliva Antigen Rapid Test Tigsun COVID-19 Speichel Antigen-Schnelltest
  Arms: Rapid antigen testing kit use once weekly; Rapid antigen testing kit use twice weekly

SUMMARY:
Our current focus is to reduce the spread of COVID through distribution of Rapid Antigen Test Kits (ATKs) to low-income, high-risk communities across Bangkok.

Hospitals across Thailand have been operating over capacity for many months, both in receiving the high number of cases as well as in testing for COVID. RT PCR, although highly sensitive, requires potentially infectious people to travel to testing sites, wait in line, and takes 1-2 days to return results, leading to further spread of COVID through increased contact with other high-risk individuals.

On the contrary, testing via an Antigen Test Kit (ATK) can be done by everyone at home with the potential to test more frequently than the PCR test due to much cheaper cost. This means that ATK testing can be mixed into people's daily lifestyle, but another underlying reason is that ATKs only show test results as positive only when an infected person is contagious. Another key advantage is the rapid results, which helps people identify risks quickly, limiting spread even faster.

Our trial therefore aims to achieve the following primary objective:

To monitor the results of freely distribute ATKs in real environments to measure its effectiveness in reducing COVID spread in communities by comparing the incidence of COVID-19 between communities with rapid antigen tests and without rapid antigen tests.

Secondary objectives are:

1. To compare the incidence of severe COVID-19 between communities with rapid antigen tests and without rapid antigen tests.
2. To study the decrease in incidence of community-acquired COVID-19 in communities with rapid antigen tests.
3. To study factors affecting community-acquired COVID-19 in these communities.
4. To campaign for the government to recognize the importance and effectiveness of weekly testing, and propose suitable strategies to fight COVID.

DETAILED DESCRIPTION:
The cluster randomized controlled trial will be conducted in Bangkok communities supported by Thaicare. A total number of 70,000 participants will be enrolled from 70 clusters. (1,000 from each cluster). Participants from each area will be divided into three groups according to the accommodation type. The rational between intervention group 1 to intervention group 2 and control group will be 1:1:1. The characteristics of population in each stratum will be reproduced as closely as possible. Cluster randomization by software will be used to blind the order of randomization. Demographic data (i.e., age, gender, weight, height, body mass index), concomitant diseases, income, type of accommodation, vaccination profile) of the control and intervention groups will be collected. The collection of data and the obtaining of the consent will be conducted by Socialgiver volunteers. There will be 2 intervention groups. Group 1 will receive 4 rapid antigen kits at the beginning of the study and will be asked to conduct a weekly self-test for 3 weeks. Group 2 will receive 7 rapid antigen kits at the beginning of the study and will be asked to conduct a twice-weekly self-test for 3 weeks (total of 6 tests)

ELIGIBILITY:
Inclusion criteria (community level): every Bangkok community under Thai Care. Exclusion criteria (community level): any Bangkok community in which the community coordinator cannot participate in the study.

Inclusion criteria (individual level): anyone who are over 10 years old. Exclusion criteria (individual level): anyone who are not consent or unable to give consents. Those who are known to be COVID-19 positive or currently treated with favipiravir

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70000 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Incidence rate of COVID19 infection | 3 week
  Incidence rate of COVID19 infection in intervention group and control group

SECONDARY OUTCOMES:
Incidence rate of severe COVID19 infection | 3 week
  severe COVID19 infection defined as ICU admission, on mechanical ventilator in intervention group and control group
Incidence of COVID19 infection in COVID19 vaccinated and non vaccinated people | 3 week
sensitivity and specificity of rapid antigen testing kit | 3 week
  compare with standard PCR

CONTACTS AND LOCATIONS:
Overall Officials: Gasit Saksirisampant, MD, Principal Investigator — Mahidol University; Dhammika Leshan Wannigama, MD.PhD, Study Chair — Chulalongkorn University; Katika Akksilp, MD, Study Director — Ministry of Health, Thailand
Locations (6):
- Thailand (6):
  - Provincial Community Housing Complex, Bangkok
  - Rural Community, Chiang Mai
  - Rural Community, Chiang Rai
  - Rural Community, Mae Hong Son
  - Rural Community, Phang Nga
  - Rural Community, Ranong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yue H, Bai X, Wang J, Yu Q, Liu W, Pu J, Wang X, Hu J, Xu D, Li X, Kang N, Li L, Lu W, Feng T, Ding L, Li X, Qi X; Gansu Provincial Medical Treatment Expert Group of COVID-19. Clinical characteristics of coronavirus disease 2019 in Gansu province, China. Ann Palliat Med. 2020 Jul;9(4):1404-1412. doi: 10.21037/apm-20-887. Epub 2020 Jul 13. PMID 32692208
- [Background] Pavelka M, Van-Zandvoort K, Abbott S, Sherratt K, Majdan M; CMMID COVID-19 working group; Institut Zdravotnych Analyz; Jarcuska P, Krajci M, Flasche S, Funk S. The impact of population-wide rapid antigen testing on SARS-CoV-2 prevalence in Slovakia. Science. 2021 May 7;372(6542):635-641. doi: 10.1126/science.abf9648. Epub 2021 Mar 23. PMID 33758017
- [Background] Hirotsu Y, Maejima M, Shibusawa M, Nagakubo Y, Hosaka K, Amemiya K, Sueki H, Hayakawa M, Mochizuki H, Tsutsui T, Kakizaki Y, Miyashita Y, Yagi S, Kojima S, Omata M. Comparison of automated SARS-CoV-2 antigen test for COVID-19 infection with quantitative RT-PCR using 313 nasopharyngeal swabs, including from seven serially followed patients. Int J Infect Dis. 2020 Oct;99:397-402. doi: 10.1016/j.ijid.2020.08.029. Epub 2020 Aug 12. PMID 32800855
- [Background] Mak GC, Cheng PK, Lau SS, Wong KK, Lau CS, Lam ET, Chan RC, Tsang DN. Evaluation of rapid antigen test for detection of SARS-CoV-2 virus. J Clin Virol. 2020 Aug;129:104500. doi: 10.1016/j.jcv.2020.104500. Epub 2020 Jun 8. PMID 32585619
- [Background] Agullo V, Fernandez-Gonzalez M, Ortiz de la Tabla V, Gonzalo-Jimenez N, Garcia JA, Masia M, Gutierrez F. Evaluation of the rapid antigen test Panbio COVID-19 in saliva and nasal swabs in a population-based point-of-care study. J Infect. 2021 May;82(5):186-230. doi: 10.1016/j.jinf.2020.12.007. Epub 2020 Dec 9. No abstract available. PMID 33309541

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT05047900/Prot_SAP_000.pdf